CLINICAL TRIAL: NCT05872633
Title: An Online Self-management Intervention for Patients With Hand Osteoarthritis - a Randomized Controlled Trial
Brief Title: Online Self-management in Hand Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Leiden University (Other)
Collaborators: Leiden University Medical Center (Other)
Responsible Party: Principal Investigator, Andrea W.M Evers, PhD, Professor, Leiden University
Organization: Leiden University Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P15.379
Record Dates: First submitted 2023-03-30; First posted 2023-05-24 (Actual); Last update posted 2023-05-24 (Actual); Status verified 2023-05

CONDITIONS: Osteoarthritis; Musculoskeletal Diseases; Rheumatic Diseases; Arthritis; Joint Diseases
Keywords: internet-based cognitive-behavioral therapy; cognitive-behavioral therapy; web-based; self-management; hand osteoarthritis
MeSH Terms: conditions — Osteoarthritis; Musculoskeletal Diseases; Rheumatic Diseases; Arthritis; Joint Diseases

STUDY DESIGN:
Masking Description: Blinding of participants and practitioners is not possible due to the nature of the study. However, the statistician who creates the randomization schedule and performs statistical analyses is blinded to group allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Online self-management intervention (and care-as-usual) (Experimental): At the start of the treatment, a face-to-face introductory meeting takes place between the participant and a psychologist, for acquaintance and to formulate goals for the treatment. Subsequently, a tailored self-management intervention, based on cognitive-behavioral therapeutic methods will be offered via an online program. Treatment will be conducted by a therapist who is specifically trained in the tailored cognitive-behavioral protocol. After finishing the online program, patients will be approached by their treating psychologist for two booster sessions via telephone. In these booster sessions it will be evaluated how the patient further attained his/her pre-set goals for the intervention. Strategies to strengthen the achieved results will be discussed. The booster sessions will take place 1 month and 2,5 months after finishing the online program.
  Interventions: Behavioral: Online self-management intervention
- Care-as-usual (Other): Care-as-usual encompasses a consultation with the rheumatologist and a 1,5-hour consultation with a clinical nurse or occupational therapist of the Leiden University Medical Center. During this consultation, patients receive information on the nature of osteoarthritis, the prognosis, and available treatment modalities, and education on chronic pain, joint protection, healthy life style, and assistive devices.
  Interventions: Other: Care-as-usual

INTERVENTIONS:
Behavioral: Online self-management intervention
  Arms: Online self-management intervention (and care-as-usual)
Other: Care-as-usual
  Arms: Care-as-usual

SUMMARY:
NB. This study has been previously registered with the National Trial Registry (NTR6266) that has been cancelled. The registered trial has been automatically transferred to a new "Landelijk Trial Register", which does not contain all correct information on the current study and where no corrections can be made. Hence, the current study has been registered again with ClinicalTrials.gov.

The goal of this clinical trial is to study the effectiveness of an online self-management intervention in adult patients with hand osteoarthritis and to explore the possibilities to implement the intervention in clinical practice after the study period. An RCT will be performed, in which 70 participants will be randomized to either care-as-usual (hand osteoarthritis care path, including consultation with the rheumatologist and a 1,5-hour consultation with a clinical nurse or occupational therapist, n=35) or care-as-usual plus the online self-management intervention (n=35). The primary effect constitutes of the difference in change in pain coping between patients in the intervention and control condition from baseline to post-intervention. As secondary outcomes, a number of other psychological and physical outcome measures will be assessed (e.g., health-related quality of life, well-being, pain impact on daily life, pain cognitions). Also, cost-effectiveness of the intervention will be measured, by assessing productivity loss and health care use of participants (using iPCQ and iMCQ).

DETAILED DESCRIPTION:
Rationale: Hand osteoarthritis has a high clinical burden, as reflected by considerable pain, decreased strength and mobility, physical disability, and an often-decreased health-related quality of life. Self-management factors related to physical and psychosocial adjustment, such as patients' perceptions about their disease and coping, play an important role in heath-related quality of life and functional ability in patients with chronic diseases, such as osteoarthritis. Improving capacities of patients in managing a chronic condition is increasingly recognized as important in the treatment of (somatic) conditions and is becoming more common in clinical practice and research. In this study, the effect of an online self-management intervention focusing on coping skills related to chronic pain in comparison to care-as-usual is studied.

Objective: To study the effectiveness of the online self-management intervention in patients with hand osteoarthritis and to explore the possibilities to implement the intervention in clinical practice after the study period.

Study design: An RCT will be performed, in which 70 participants will be randomized to either care-as-usual (hand osteoarthritis care path, including consultation with the rheumatologist and a 1,5-hour consultation with a clinical nurse or occupational therapist, n=35) or care-as-usual plus the online self-management intervention (n=35). Baseline, post-intervention, 6-week, and three-month follow-up questionnaires will be used to measure primary and secondary outcomes. To assess implementation possibilities of the online intervention, structured qualitative interviews among patients and health professionals will examine to what extent the intervention suits the needs and skills of patients and to what extent the intervention fits within the current care process.

Study population: All patients ≥18 years with hand osteoarthritis who are referred to the hand osteoarthritis care path at the rheumatology clinic at Leiden University Medical Center with on-going pain complaints during at least three months will be invited to participate in the study. Patients need to be fluent in Dutch, need to be able to give informed consent, and have internet access. Severe psychiatric co-morbidity, on-going psychological treatment elsewhere, difficulties with (written) communication, a lack of internet literacy, and having secondary osteoarthritis are exclusion criteria.

Intervention: The intervention is based on cognitive-behavioral methods. It starts off with a face-to-face introduction consultation. Subsequently, the tailored self- management intervention will be offered via an online program. The intervention consists of six modules containing pain education, practical assignments, relaxation training, and registrations. The first and last modules are an introductory and closure module; in between are four modules aimed at learning how to cope with the consequences of a chronic condition in daily life. The modules focus on (1) activity, (2) mood, (3) thoughts, and (4) the social environment. At least once a week, participants receive feedback on the assignments and motivational support from a psychologist, by means of text messages in a secured mail box in the online program. After finishing the online program, patients will be approached by their treating psychologist for two booster sessions via telephone. In these booster sessions it will be evaluated how the patient further attained his/her pre-set goals for the intervention. Strategies to strengthen the achieved results will be discussed. The booster sessions will take place 1 month and 2,5 months after finishing the online program.

Main study parameters/endpoints: The primary effect constitutes of the difference in change in pain coping between patients in the intervention and control condition from baseline to post-intervention. As secondary outcomes, a number of other psychological and physical outcome measures will be assessed (e.g., health-related quality of life, well-being, pain impact on daily life, pain cognitions). Also, cost-effectiveness of the intervention will be measured, by assessing productivity loss and health care use of participants (using iPCQ and iMCQ).

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: In the control group the usual standard of care is provided. In the intervention group patients will be offered an internet-based self-management intervention, which potentially improves their pain coping and other psychological and physical outcomes. No risk is involved with participation in this study. The only burden for participants is investment of time.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with hand osteoarthritis, following American College of Rheumatology (ARC) criteria (Altman et al., 1990)
* Referred to the hand osteoarthritis care path
* Complaints from hand osteoarthritis including pain, with a minimal duration of 3 months
* Minimum age of 18 years
* Fluent in Dutch language
* Able to give informed consent
* Own a computer with internet access

Exclusion Criteria:

* Difficulties with (written) communication (e.g., due to analphabetism) and lack of internet literacy
* Severe psychiatric comorbidities that interfere with the study protocol
* On-going psychological treatment elsewhere
* Patients with secondary osteoarthritis due to diseases, such as 1) inflammatory rheumatic diseases, such as rheumatoid arthritis, psoriatic arthritis, etc., 2) bone diseases, such as M. Paget, osteochondritis, 3) metabolic diseases associated with joint disease, such as hemochromatosis, acromegaly, 4) severe crystal arthropathies, such as tophaceous polyarticular gout.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2016-08-01 (Actual); Primary Completion 2021-05-19 (Actual); Study Completion 2021-05-19 (Actual)

PRIMARY OUTCOMES:
Change in pain coping | Baseline, immediately after the intervention, at 6 weeks and 3 months follow-up.
  A visual analogue scale (VAS) from 0 to 10 will be used to assess pain coping, with higher scores indicating better pain coping. The primary endpoint is the difference in change in pain coping between patients in the intervention and control condition from baseline to post-intervention (immediately after the intervention).

SECONDARY OUTCOMES:
Change in well-being | Baseline, immediately after the intervention, at 6 weeks and 3 months follow-up.
  A VAS from 0 to 10 will be used to assess well-being, with higher scores indicating better well-being.
Change in illness cognitions | Baseline, immediately after the intervention, at 6 weeks and 3 months follow-up.
  Illness cognitions will be measured by the Illness Cognition Questionnaire (ICQ) (specifically, Helplessness and Acceptance scales). Items are scored on a 4-point Likert scale ranging from "not at all" to "completely". Higher scale scores indicate greater use of the measured construct.
Change in pain coping strategies | Baseline, immediately after the intervention, at 6 weeks and 3 months follow-up.
  Pain coping strategies will be measured by the Pain Coping Inventory (PCI). The questionnaire consists of six scales; Pain Transformation, Distraction, and Reducing Demands are characterized as active pain coping strategies, and Retreating, Worrying, and Resting are classified as passive pain coping strategies. Items are scored on a 4-point Likert scale ranging from "hardly ever" to "very often", with higher scale scores indicate greater use of the measured coping strategy.
Change in illness perceptions | Baseline, immediately after the intervention, at 6 weeks and 3 months follow-up.
  Illness perceptions will be measured by the Illness Perception Questionnaire (IPQ-R). The Identity scale consists of the sum of yes-rated items (whether patients believe certain symptoms to be related to their illness). Furthermore, the Timeline Acute/Chronic, Timeline Cyclical, Consequences, Illness Coherence, Personal Control, Treatment Control, and Emotional Representations scales are rated on a 5-point Likert type scale ranging from "strongly disagree" to "strongly agree". High scores on the Identity, Timeline Acute/Chronic and Cyclical, Consequences, and Emotional Representations scales reflect beliefs about the number of symptoms attributed to the illness, the chronicity and cyclical nature, and the negative consequences of the illness, and patients' emotional experience of their illness. High scores on the Personal and Treatment Control and Coherence scales reflect positive beliefs about perceived control and an understanding of the illness.
Change in pain | Baseline, immediately after the intervention, at 6 weeks and 3 months follow-up.
  A VAS from 0 to 10 will be used to assess pain, with higher scores indicating more severe pain.
Change in pain and disability | Baseline, immediately after the intervention, at 6 weeks and 3 months follow-up.
  The Pain and Disability scales will be used of the Australian/Canadian Hand Osteoarthritis Index (AUSCAN). Items are rated on 5-point Likert scale ranging from "none" to "extreme", with higher scores indicating more pain and disability.
Change in pain interference in daily functioning and pain severity, and as exploratory measures support, life control, and affective distress | Baseline, immediately after the intervention, at 6 weeks and 3 months follow-up.
  Part 1 of the Multidimensional Pain Inventory-Dutch Language Version (MPI-DLV) will be used, with the scales Interference and Pain Severity, and as exploratory measures Support, Life Control, and Affective Distress. Items are rated on various 7-point Likert scales, with higher scores indicating greater intensity in a subscale.
Change in health-related quality of life | Baseline, immediately after the intervention, at 6 weeks and 3 months follow-up.
  Health-related quality of life will be measured by the RAND-36, which comprises 36 items that are averaged together to provide eight health scale scores, namely Physical Functioning, Role Limitations due to Physical Health Problems, Role Limitations due to Personal or Emotional Problems, Social Functioning, Emotional Well-being, Energy/Fatigue, Bodily Pain, and General Health Perceptions. It also includes one item on perceived change in health. Moreover, physical and mental health composite scores will be calculated. Higher scores indicate more advantageous health states.
Change in health-related quality of life | Baseline, immediately after the intervention, at 3 months follow-up.
  Health-related quality of life will be measured by the the Five-Level Version of the EQ-5D (EQ-5D-5L). Five dimensions are assessed in 5 items: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. A 5-point Likert scale ranging from "no problems" to "extreme problems" is applied, with higher scores corresponding with more problems in a HR-QoL dimension. Moreover, a VAS from 0 to 100 (0 = "The best health you can imagine" to 100 = "The worst health you can imagine") is used, with higher scores indicating a better perceived health state.

OTHER OUTCOMES:
Economic evaluation: Five-Level Version of the EQ-5D (EQ-5D-5L) | Baseline, immediately after the intervention, at 3 months follow-up.
  The intervention will be economically evaluated using the Five-Level Version of the EQ-5D (EQ-5D-5L). Five dimensions are assessed in 5 items: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. A 5-point Likert scale ranging from "no problems" to "extreme problems" is applied, with higher scores corresponding with more problems in a HR-QoL dimension. The 5 dimensions can be summed into a health state. Utility values can be calculated for these health states.
Economic evaluation: iMTA Medical Consumption Questionnaire (iMCQ) | Baseline, immediately after the intervention, at 3 months follow-up.
  The intervention will be economically evaluated using the iMTA Medical Consumption Questionnaire (iMCQ). The iMCQ measures health-care utilization.
Economic evaluation: iMTA Productivity Cost Questionnaire (iPCQ) | Baseline, immediately after the intervention, at 3 months follow-up.
  The intervention will be economically evaluated using the iMTA Productivity Cost Questionnaire (iPCQ). In this questionnaire, productivity losses are measured in three modules, so that specific types of productivity losses can be left out when these are not applicable to a specific population.
Patient satisfaction | Immediately after the intervention.
  After the intervention period, patient satisfaction and experience with the intervention, and perceived effect of the intervention will be evaluated with an evaluation questionnaire consisting of various numerical rating scales, Likert scales and open questions.
Expected/perceived patient-provider interaction | Baseline and immediately after the intervention.
  The expected/perceived patient-provider interaction will be measured with the Internet-specific Therapeutic Relationship Questionnaire (ITRQ). The ITRQ consists of 10 items rated on a 10-point Likert scale ranging from "totally disagree" to "completely agree". It comprises two scales (Internet-specific Time and Attention and Internet-specific Reflection and Comfort) and a total score. Higher scores indicate a stronger therapeutic relationship.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Evers, PhD, Principal Investigator — Leiden University

IPD SHARING:
Plan to Share IPD: Yes
Once an article on the study is published, a publication package will be published on DataverseNL. This package includes the manuscript, procedures, raw data files, computer code, and processed data files.
Supporting Information: SAP
Time Frame: IPD will become available once an article on the study is published on DataverseNL; the statistical analysis plan will be published on ClinicalTrials.gov during registration (before data analysis takes place).
Access Criteria: Open access.

REFERENCES:
- [Derived] Terpstra JA, van Beugen S, van der Vaart R, van Eersel RA, Dusseldorp E, Kloppenburg M, Evers AWM. An internet-based cognitive-behavioral self-management intervention for patients with hand osteoarthritis or fibromyalgia - Two randomized controlled trials. Internet Interv. 2026 Jan 19;43:100908. doi: 10.1016/j.invent.2026.100908. eCollection 2026 Mar. PMID 41631249

DOCUMENTS (1):
  • Statistical Analysis Plan (2022-07-25): https://cdn.clinicaltrials.gov/large-docs/33/NCT05872633/SAP_000.pdf